CLINICAL TRIAL: NCT04358120
Title: A Multicentre Clinical Investigation to Assess Efficacy and Safety of Intra-articular Injections of a New Viscosupplement Based on Hyaluronic Acid Combined With Chondroitin Sulfate in Patients With Knee Osteoarthritis
Brief Title: A Multicentre Clinical Investigation to Assess Efficacy and Safety of Intra-articular Injections of Hyaluronic Acid Combined With Chondroitin Sulfate in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RR82-17-01
Record Dates: First submitted 2020-03-02; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-03

CONDITIONS: Osteo Arthritis Knee
Keywords: Hyaluronic Acid; Chondroitin sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyaluronic Acid Combined With Chondroitin Sulfate (Other): The treatment consists of 3 intra articular injections of Hyaluronic Acid With Chondroitin Sulfate administered one per week for 3 consecutive weeks: the 1st at Visit 1 (Week 0), the 2nd at Visit 2 (Week 1) and the 3rd at Visit 3 (Week 2)
  Interventions: Device: Hyaluronic Acid Combined With Chondroitin Sulfate

INTERVENTIONS:
Device: Hyaluronic Acid Combined With Chondroitin Sulfate — Subjects' participation in the study will last 26 weeks. The study includes 7 visits that consist of a Screening visit, three treatment visits and three follow-up visits.
  Eligible subjects will undergo a Baseline visit (V1 at week 0) during which, after the confirmation of eligibility, assessments and ultrasound evaluation, the study subjects will be treated with the 1st injection of 2%Hyaluronic Acid and 2% chondroitin sulfate Subsequent treatments will be administered at weekly intervals during Visit 2 (V2 at week 1) and Visit 3 (Visit 3 at week 2) after the effectiveness assessments.
  Study subjects will return for Follow-up visits 1 month (Visit 4 at week 6), 3 months (Visit 5 at week 14) and 6 months (Visit 6 at week 26) after the last injection

SUMMARY:
This is a multicentre, prospective, sponsor initiated clinical investigation that aims to evaluate safety and efficacy of Hyaluronic Acid Combined With Chondroitin Sulfate in symptomatic patients with OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* At Screening

  * Male or female between the ages of 40 and 80
  * Body Mass Index (BMI) ≤ 30;
  * Mean knee pain score at rest over the last 24 hours evaluated on VAS (0-100) ≥ 40. The most painful knee is considered the target knee;
  * OA of the Knee radiologically and clinically confirmed responding to criteria of American College of Rheumatology (ACR): pain of the knee and crepitus on active motion or morning stiffness less than 30 minutes or age >50 years
  * Symptomatic knee pain for more than 6 months;
  * Radiological Kellgren and Lawrence grade II or III confirmed by an X-ray not older than 12 months;
  * Willing to discontinue any systemic analgesic/NSAID therapy, opioids, systemic corticosteroids, skeletal muscle relaxants, and any other medication that would interfere with the study assessments, except for the rescue medication, with no intention to resume them during the clinical investigation (see Appendix 5 for wash out period);
  * Patient able to comply with the instructions of the clinical investigation and to maintain a Rescue Medication Diary during the study;
  * Having signed the study informed consent.
* at Baseline

  * Patient does not have chondromatosis or villonodular synovitis of the knee evaluated by Ultrasound;
  * Patient has complied with the requirements for rescue medication (no more than 6 tablets or 3 grams of paracetamol per day up to 4 days per week and paracetamol discontinued 24 hours before first IA injection);
  * Mean knee pain score at rest over the last 24 hours evaluated on VAS (0 - 100) ≥ 40 (with a washout period for Paracetamol of 24 hours);
  * Patient has discontinued prior to Baseline the use of all prohibited medications in accordance with the washout period defined in Appendix 5;
  * Patient continues to meet all Screening inclusion/exclusion criteria at the Baseline visit.

Exclusion Criteria:

* Related to the OA pathology

  * Recent trauma (< 1 month) of the target knee responsible for the symptomatic knee pain;
  * Articular disease resulting from articular dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, haemophilia, hemochromatosis;
  * Inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, gout and infectious arthritis, acute calcium pyrophosphate arthritis);
  * Pathologies interfering with the evaluation of OA. Related to treatments
  * Corticosteroids injection in the target knee in the last 3 months before first intra-articular (IA) injection;
  * Hyaluronan injection in the target knee in the last 6 months before first IA injection;
  * Arthroscopy and surgery in the target knee in the last 3 months before first IA injection;
  * Oral corticosteroid therapy ≥ 5mg/day (in Prednisone equivalent) in the last 3 months before first IA injection;
  * OA treatments based on curcuma extract in the last 3 months before first IA injection;
  * Change in the dosage of symptomatic slow-acting drugs (SYSADOA) e.g., chondroitin, glucosamine, diacerein or avocado-soya unsaponifiables in the last 3 months before first IA injection;
  * Contraindications to 4% GAG: hypersensitivity to the product components;
  * Infections or skin diseases in the area of the injection site;
  * Change in the dosage of ongoing non-pharmacologic therapy for the lower extremities (including physical therapy) initiated in the month before first injection;
  * Anticoagulant (coumarinic compound) and heparin. Related to associated diseases
  * Severe diseases (e.g., liver or renal failure, lung/heart disease, tumour, HIV);
  * Severe alteration of mobility interfering with the functional evaluation;
  * High risk of haemorrhage;
  * Patient with known allergy to paracetamol;
  * Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee.

Related to study subjects

* Participation to a therapeutic clinical trial in the last 3 months before first injection;
* Pregnancy, breastfeeding, planned conception and premenopausal women without contraception, tubal ligation or hysterectomy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Change in pain score measured by Visual Analogue Scale (VAS) | at week 6, 14 and 26
  Change in pain perception from baseline in patient with knee osteoarthritis after three intra-articular 2% Chondroitin Sulfate + 2% hyaluronic Acid injections assessed by Visual Analogue Scale (VAS) (From 0 to 100) at weeks 6, 14 and 26

SECONDARY OUTCOMES:
Change in Patient's Global Assessment | at weeks 6, 14 and 26
  Change from baseline up to 26 weeks after first treatment in Patient's Global Assessment of knee functional disability, assessed by VAS (0-100)
Change from baseline in knee pain and function up to 26 weeks | at weeks 6, 14 and 26
  Change from baseline provided by the intra-articular 2% Chondroitin Sulfate + 2% Hyaluronic Acid injections measured by Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index (0-100 mm) for knee at weeks 6, 14 and 26
Change from baseline up to 26 weeks after first treatment on knee functional disability on Clinical Observer Global Assessment (COGA) | at weeks 6, 14 and 26
  Change from baseline up to 26 weeks after first treatment in COGA of knee functional disability, assessed by VAS (0-100)
Number of patients Responder to treatment | Weeks 6, 14 and 26
  Number of patients with clinical response to treatment using the OMERACT-OARSI set of criteria: high improvement in pain or function ≥ 50% or improvement in at least 2 of the 3 of the following criteria: high improvement in pain or function ≥ 50% or improvement in at least 2 of the 3 following:
  * pain ≥ 20% and absolute change ≥10,
  * function ≥20% and absolute change ≥10,
  * PGA ≥ 20% and absolute change ≥10.
Change from baseline in Synovitis at 6 weeks | at week 6
  Change in Synovitis at week 6 vs week 0 assessed by ultrasound scored according to the scoring systems proposed by OMERACT US on knee OA.
  A global score for synovitis corresponds to the maximum score for synovitis obtained at the suprapatellar or parapatellar recesses.
  Synovitis (grades 0-3): Grade 0 = no synovitis, Grade 1= minimal distension, Grade 2= moderate distension or enlargement, Grade 3= severe distension or enlargement of the recess
Change from baseline in Synovial hypertrophy at 6 weeks | at week 6
  Change in Synovial hypertrophy at week 6 vs week 0 assessed by ultrasound scored according to the scoring systems proposed by OMERACT US on knee OA.
  Synovial hypertrophy (0-1) where 0= absence, 1= presence
Change from baseline in knee Effusion at 6 weeks | at week 6
  Change in Effusion at week 6 vs week 0 assessed by ultrasound scored according to the scoring systems proposed by OMERACT US on knee OA.
  Effusion (0-1) 0= absence, 1= presence
Change from baseline in popliteal cyst at 6 weeks | at week 6
  Change in Popliteal cyst at week 6 vs week 0 assessed by ultrasound scored according to the scoring systems proposed by OMERACT US on knee OA.
  Popliteal cyst (0-1) 0= absence, 1= presence
Change in Synovial Power Doppler signal at week 6 | at week 6
  Changein Synovial Power Doppler signal at week 6 vs week 0 assessed by ultrasound.
  Synovial Power Doppler signal (0-1) and (0-3) Grade 0 = no intra-articular colour signal Grade 1 = up to three signal colour signals or two single and one confluent colour signals representing only low flow
Safety of the treatment. Number of patient with treatment related adverse events | through study completion
  Safety evaluation by tracking the number of patient withdrawals and their adverse events correlated to treatment at each visit

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (5):
  - Revmacentrum MUDr. Mostera,, Brno
  - Rheumatology, Polyclinic Lesná, Brno
  - Institute of rheumatology, Prague
  - University Hospital Motol, Department of Rheumatology of Children and Adults, Prague
  - Medical Plus, s.r.o, Uherské Hradiště